CLINICAL TRIAL: NCT02409121
Title: A Novel Health Information Technology System (BMT Roadmap) for Pediatric BMT Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2015.050; HUM00100126 (Other: University of Michigan)
Record Dates: First submitted 2015-03-27; First posted 2015-04-06 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Leukemia; Lymphoma; Brain Tumor
Keywords: hematopoietic cell transplantation; caregivers; health information technology; patient-centered care
MeSH Terms: conditions — Leukemia; Lymphoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): All participants will receive a tablet educational intervention (health IT platform) during the patient inpatient hospitalization for autologous or allogeneic transplant
  Interventions: Behavioral: Education information system

INTERVENTIONS:
Behavioral: Education information system — Participants will receive a mobile tablet as an educational intervention during the patient's inpatient hospitalization

SUMMARY:
Hematopoietic cell transplantation (BMT), or commonly referred to as blood and marrow transplantation (BMT), is a potentially life-saving therapy for many malignant and non-malignant conditions. Despite advances over the past decade, which have led to improved outcomes, BMT remains an intense treatment modality often requiring prolonged inpatient-based care. While many patients endure the acute complications of the procedure, it is common for BMT patients and their caregivers to experience increased risk of financial and emotional burden, hospital readmission, and health service utilization. This highlights the importance of active involvement of BMT patients in their own health care (self-efficacy). For pediatric BMT patients, parents are the primary caregivers. As such, parental activation on behalf of the child (patient) plays a critical role in effective patient-parent-provider partnerships, which is increasingly recognized as the optimal model for health care delivery, particularly for those facing life-altering medical treatments. It is essential to develop effective strategies to enhance this partnership. Health information technology (IT)-mediated tools offer the potential to overcome constraints in health care delivery limited by provider time, complicated health information, and financial pressures. Significant gaps in knowledge exist on the use of health IT tools using low-cost and well-accepted delivery platforms in routine inpatient care, especially for high-risk or critically ill populations. The investigators hypothesize that a tablet-based tool displaying personal health information could provide a platform to promote caregiver (parent) activation and enhance health communication. In this clinical research study, the investigators will conduct a pilot study of an educational health IT system developed on a tablet (Apple iPad®) that the investigators refer to as a Personalized Engagement Tool (PET) or the "BMT Roadmap." The Apple iPad® was selected as the platform for delivery of the educational intervention given its ergonomic features. The implementation and evaluation of the BMT Roadmap information system in caregivers of children undergoing BMT have been based on the generation of user (caregivers and patients) needs that incorporated well-established user-centered design processes including qualitative and quantitative research methods (published and unpublished data). The assembled investigators represent a strong multidisciplinary team with complementary and integrated expertise who are well-poised to carry out the proposed research. The Protocol or Study Team includes pediatric BMT physicians, Center for Health Communications Research (CHCR) staff, health informaticist, biostatistician, and psychologist. This research study is innovative because it addresses a gap in the literature on the role of health IT in parent activation on behalf of the child in the inpatient setting of a high-risk BMT population. The BMT Roadmap information system provides a robust experimental framework for further testing the utility of other care components that relate to parent activation or participation and for potential adoption in other complex medical conditions. The new knowledge gained herein will thus contribute to the evidence base of how health IT improves health care quality and provide the basis of further study in a full-scale clinical trial.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS Title A Pilot Study of Patient and Caregiver Participation through an Educational Health Information Technology System ("The BMT Roadmap") in the Context of Hematopoietic Cell Transplantation

Objective To evaluate the usefulness and usability of a health information technology (IT) system ("The BMT Roadmap"). This educational system will be developed on an Apple iPad® with collaborators from the School of Information, Health Informatics, and the Center for Health Communications Research (CHCR). The BMT Roadmap will be used by caregivers of patients hospitalized for first-time autologous (self) or allogeneic (alternative donor) blood and marrow transplantation (BMT) as well as patients (age 10 years or older) who are hospitalized for first time autologous or allogeneic BMT. The investigators hypothesize that parents will use the BMT Roadmap to become more active participants on behalf of their child.

The information system will consist of 5 modules personalized to the study participant's child: (1) laboratory studies, (2) medications, (3) clinical trials enrolled on, (4) health care providers (BMT physicians, 7 Mott Nurses, BMT NPs, coordinators, pharmacists, nutritionist, social worker), and (5) criteria for discharge.

Sample Size Caregivers: The investigators aim to enroll 10 adult caregivers of patients (0-25 years of age) undergoing autologous (self) or allogeneic BMT (alternative donor); and Patients: 10 patients (10 years of age or older) undergoing autologous or allogeneic BMT. This sample size was determined based on the patient demographics of the University of Michigan Pediatric BMT Program. The number of participants who meet eligibility is approximately 50 per year. The investigators plan to enroll approximately 2 adult caregivers and 2 patients per month for an estimated accrual time of 5 months. This study allows for concurrent enrollment in other trials.

Study Design After signing an informed consent, participants will be provided with an Apple iPad®. Qualitative and quantitative research methods will be used to measure the study outcomes. There will be approximately 6-8 qualitative interviews per participant conducted periodically from pre-BMT until 100 days post-BMT. Additionally, 15-20 qualitative interviews will be conducted of BMT care providers, including physicians, nurses, pharmacists, nutritionists, social worker, and psychologist to evaluate their attitudes and perceptions of the BMT Roadmap information system. Quantitative survey instruments will only be administered to adult participants (age 18 years or older). Caregivers with children (patients) who are younger than 10 years of age may be eligible to participate even though their children are too young to assent or participate themselves.

Inclusion Criteria Caregivers: Caregiver (age 18 years or older) of a patient (0-25 years of age) who is an inpatient undergoing autologous or allogeneic BMT; Patients: patient (10 years or older) who is inpatient undergoing autologous or allogeneic BMT. Ability to speak and read proficiently in English (the study's instruments have not been translated and validated in languages other than English); Willing and able to provide informed consent; Willing to comply with study procedures and reporting requirements.

Treatment Plan This protocol is an educational intervention study (no more than minimal risk). It does not include treatment of an investigation agent treatment.

Study Endpoints The primary outcome measures will be the usefulness and the usability of the BMT Roadmap information system. Secondary measures will include standard-of-care patient-related clinical outcomes (length of stay and risk of day 30 and 100 readmission, infections, transplant-related mortality, and survival).

Data Analysis Descriptive statistics will be calculated for each survey instrument. Univariate analyses will be performed to assess associations between the instruments and demographic, social, and environmental characteristics of the parent (type of insurance, marital status, number of children in household), and disease-related characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited by BMT RN Coordinators and physicians prior to patient admission to the Pediatric BMT Unit. Caregiver (age 18 years or older) of any patient eligible to undergo autologous or allogeneic BMT and any patient (age 10 years or older) eligible to undergo autologous or allogeneic BMT will be recruited during the "Pre-Transplant Work-up" stage in the outpatient setting.
* CAREGIVER PARTICIPANTS: Caregiver (age 18 years or older) of a patient who will be hospitalized to undergo first-time autologous (self) or allogeneic (alternative donor) BMT in the University of Michigan Mott Children's Hospital Pediatric BMT Unit. The age range of patients typically transplanted in the Pediatric BMT unit is 0-25 years. Caregivers with children (patients) who are younger than 10 years of age may be eligible to participate even though their children are too young to assent or participate themselves.
* PATIENT PARTICIPANTS: Patient (age 10 years or older) who will be hospitalized to undergo first-time autologous or allogeneic BMT will be given the opportunity to assent/consent and participate in the study. With his/her permission, the patient will also be provided with their own iPad® BMT Roadmap information system to use. Qualitative interviews will be conducted in patients (age 10 years or older) with their assent/consent. However, patients (age 10-17.9 years) will not be asked to complete surveys, because they have not been validated in this age group. Patients (18 years or older) will be asked to complete surveys. The upper age limit is typically 25 years on the Pediatric BMT Unit. This limit will be determined by only those patients undergoing transplant in the Pediatric BMT Unit.
* Ability to speak and read proficiently in English (the study's instruments have not been translated and validated in languages other than English)
* Willing and able to provide informed consent
* Willing to comply with study procedures and reporting requirements.

Exclusion Criteria:

* Not willing and able to provide informed consent.
* Not willing to comply with study procedures and reporting requirements.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects who participate in the health information technology educational intervention | 100 days
  feasibility of recruitment and retention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Fauer AJ, Hoodin F, Lalonde L, Errickson J, Runaas L, Churay T, Seyedsalehi S, Warfield C, Chappell G, Brookshire K, Chaar D, Shin JY, Byrd M, Magenau J, Hanauer DA, Choi SW. Impact of a health information technology tool addressing information needs of caregivers of adult and pediatric hematopoietic stem cell transplantation patients. Support Care Cancer. 2019 Jun;27(6):2103-2112. doi: 10.1007/s00520-018-4450-4. Epub 2018 Sep 20. PMID 30232587
- [Derived] Maher M, Kaziunas E, Ackerman M, Derry H, Forringer R, Miller K, O'Reilly D, An LC, Tewari M, Hanauer DA, Choi SW. User-Centered Design Groups to Engage Patients and Caregivers with a Personalized Health Information Technology Tool. Biol Blood Marrow Transplant. 2016 Feb;22(2):349-358. doi: 10.1016/j.bbmt.2015.08.032. Epub 2015 Sep 5. PMID 26343948